CLINICAL TRIAL: NCT04648423
Title: Multinational, Multicentre, Double-blind, Placebo-controlled Evaluation of the Efficacy of GHB in the Long-term Maintenance of Abstinence in Alcoholic Patients After the Initial Weaning Phase, Stratified by Lesch's Taxonomy (GATE 2)
Brief Title: Evaluation of the Efficacy of Sodium Oxybate in the Long-term Maintenance of Abstinence in Alcoholic Patients
Acronym: GATE2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorio Farmaceutico Ct S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHBCR00/2
Record Dates: First submitted 2020-11-16; First posted 2020-12-01 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Alcohol Use Disorder (AUD); Alcohol Dependence
Keywords: alcoholism; alcohol; alcohol dependence; relapse prevention
MeSH Terms: conditions — Alcoholism | interventions — Sodium Oxybate

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled study with parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The control medication (placebo) was identically-looking and identically tasting as active.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium oxybate (Experimental): Sodium oxybate solution for oral administration (175 mg/mL). Dose (body weight ≤ 65 kg): 19.0 mL daily, in 3 administrations, for 6 months Dose (body weight > 65 kg): 22.5 mL daily, in 3 administrations, for 6 months
  Interventions: Drug: Sodium Oxybate
- placebo (Placebo Comparator): Placebo solution for oral administration. Dose (body weight ≤ 65 kg): 19.0 mL daily, in 3 administrations, for 6 months Dose (body weight > 65 kg): 22.5 mL daily, in 3 administrations, for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Oxybate — solution for oral administration
  Other Names: gamma-hydroxy butyrate (GHB)
  Arms: sodium oxybate
Drug: Placebo — solution for oral administration
  Arms: placebo

SUMMARY:
Additional pharmacotherapies in the treatment of alcohol dependence are needed. Sodium oxybate showed efficacy in the maintenance of abstinence in alcohol-dependent patients in several small randomized trials of short duration. The aim of the present phase III/IV study is to confirm in a randomized-controlled study the efficacy and safety of oral sodium oxybate in the maintenance of abstinence.

DETAILED DESCRIPTION:
Alcohol dependence (AD) is the most severe form of alcohol use disorder. It occurs in 2.6% of people aged 15+ years worldwide and can result in a reduction of life-expectancy by several years as compared with the general population.

Currently, disulfiram, acamprosate and naltrexone are the main medicinal products registered for the maintenance of abstinence in AD patients. Although effective on the group level, effects sizes are limited, and many AD patients fail to respond to these medications. Therefore, additional pharmacological treatments are needed.

Sodium oxybate 50mg/kg/day showed evidence of efficacy compared to placebo and naltrexone in the maintenance of abstinence in AD patients in a series of open label and blinded randomized controlled trials (RCTs). However, studies were generally small and did not investigate the sustainability of the Sodium oxybate effect post-treatment.

The present phase III/IV RCT (GATE 2) aimed to confirm the efficacy and safety of oral Sodium oxybate in the maintenance of abstinence. Secondary aims included the assessment of sustained SMO effects during the 6-month medication free period immediately following the 6-month treatment period and monitoring the risk of Sodium oxybate dependence.

ELIGIBILITY:
Inclusion Criteria:

The following subjects were recruited:

* males and females;
* of any ethnic group;
* age between 21 and 75 years at recruitment;
* documented alcohol dependency before weaning detected according to the CAGE instrument, classified according to the DSM-IV and ICD-10 and severity rated according to the MALT instrument;
* classified according to Lesch typology;
* having successfully undergone a detoxification program, encompassing a 10-day treatment period and a subsequent 10-day untreated follow-up;
* with a responsible relative or caregiver;
* having issued the informed consent.

Exclusion Criteria:

* subjects who did not quit alcohol drinking after the detoxification period;
* subjects with history of epilepsy or epileptics seizures not properly controlled by established anti-epileptic treatment;
* subjects with dependence from narcotics or other drugs of abuse;
* subjects without a stable address;
* subjects without a reference relative or caregiver;
* subjects with renai failure (blood creatinine >2.5 mg/dL and/or documented proteinuria >500 mg/day);
* subjects with heart failure or severe respiratory failure;
* subjects with hepatic encephalopathy stage lI-IV;
* subjects with severe psychiatric disorders requiring treatment with psychoactive medications (excluding short-term benzodiazepine treatments);
* subjects under treatment with clonidine, disulfiram (after the end of the detoxification period), haloperidol, bromocryptine, serotonine re-uptake inhibitors or other serotoninergic agents;
* female subjects who cannot assure not to become pregnant during the 7-month period covering treatment and the first treatment-free month of follow-up;
* documented pre-existent hypersensitivity to GHB;
* subjects unable or unwilling to issue the informed consent;
* participating to another clinica! investigation in the previous month prior to recruitment; 15. any other medicai condition which, according to the investigator, justifies the patient's exclusion from the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2001-07-23 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Cumulative Abstinence Duration (CAD) | 6-month treatment period
  to demonstrate that sodium oxybate is superior to placebo in the CAD during the treatment period.

SECONDARY OUTCOMES:
CAD stratified | 6-month treatment period
  CAD during treatment period according to subtype patients stratified by Lesch's categories.
Assessment of the exposure-corrected CAD | 6-month treatment period
  assessment of the exposure-corrected cumulative abstinence duration (CCAD) during treatment.
CAD during the whole study | 12 months: 6-month treatment period + 6-month follow-up
  CAD during the whole observation period
Proportion of abstinent patients | 12 months: 6-month treatment period + 6-month follow-up
  proportion of abstinent patients at the end of the 6-month treatment period and at the end of the entire observation period.
Time to the first relapse | 6-month treatment period
  assessment of the time to the first relapse during the treatment period.
Change from baseline in the craving for alcohol intensity and frequency by the Lubecker Craving Risiko Ruckfall (LCRR) questionnaire. | 12 months: 6-month treatment period + 6-month follow-up
  The LCRR provides the patient's current state about his craving for alcohol. The clinician interviews the patient to rate the intensity of the desire for alcohol (item-1) on a 4-point scale ranging from 1 (no desire) to 4 (very strong desire), and to rate the frequency of the desire for alcohol (item-2) on a 6-point scale ranging from 1 (never) to 6 (nearly continuous).
  Higher scores mean a worse outcome.
Assessment of the time course of γ-GT as biological marker of alcohol abuse, during treatment and at the end of follow-up. | Month 6
  γ-GT values
Adverse events | 6-month treatment period
  evaluation of the frequency, nature and severity of adverse clinical events, including mortality and morbidity
Number of participants with Adverse Events (AEs) | 6-month treatment period
  Overview of AEs.
Risk of Secondary Dependence - treatment period | 6-month treatment period
  Evaluation of the risk of onset of dependence from the medication, by means of a 2-item questionnaire. The first to rate the intensity of the desire for medication since the last visit in a scale ranging from 0 to 100. The second to rate the approach to the next dose in a scale ranging from 1 (I just waited for the time to come) to 6 (I took the dose sooner than planned).
  Higher scores mean a worse outcome.
Assessment of the time course of MCV as biological marker of alcohol abuse, during treatment and at the end of follow-up. | Month 6
  MCV values

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cacciaglia, Study Chair — Laboratorio Farmaceutico C.T.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Skala K, Caputo F, Mirijello A, Vassallo G, Antonelli M, Ferrulli A, Walter H, Lesch O, Addolorato G. Sodium oxybate in the treatment of alcohol dependence: from the alcohol withdrawal syndrome to the alcohol relapse prevention. Expert Opin Pharmacother. 2014 Feb;15(2):245-57. doi: 10.1517/14656566.2014.863278. Epub 2013 Nov 28. PMID 24283802
- [Result] van den Brink W, Addolorato G, Aubin HJ, Benyamina A, Caputo F, Dematteis M, Gual A, Lesch OM, Mann K, Maremmani I, Nutt D, Paille F, Perney P, Rehm J, Reynaud M, Simon N, Soderpalm B, Sommer WH, Walter H, Spanagel R. Efficacy and safety of sodium oxybate in alcohol-dependent patients with a very high drinking risk level. Addict Biol. 2018 Jul;23(4):969-986. doi: 10.1111/adb.12645. PMID 30043457
- [Derived] Guiraud J, Addolorato G, Antonelli M, Aubin HJ, de Bejczy A, Benyamina A, Cacciaglia R, Caputo F, Dematteis M, Ferrulli A, Goudriaan AE, Gual A, Lesch OM, Maremmani I, Mirijello A, Nutt DJ, Paille F, Perney P, Poulnais R, Raffaillac Q, Rehm J, Rolland B, Rotondo C, Scherrer B, Simon N, Skala K, Soderpalm B, Somaini L, Sommer WH, Spanagel R, Vassallo GA, Walter H, van den Brink W. Sodium oxybate for the maintenance of abstinence in alcohol-dependent patients: An international, multicenter, randomized, double-blind, placebo-controlled trial. J Psychopharmacol. 2022 Oct;36(10):1136-1145. doi: 10.1177/02698811221104063. Epub 2022 Jul 7. PMID 35796481